CLINICAL TRIAL: NCT02951494
Title: Einfluss Der Körpergewichtsunterstützung Auf Einem AlterG®-Antigravitationslaufband Auf Die Kardiopulmonale Leistungsfähigkeit Und Trainierbarkeit
Brief Title: Impact of Lower Body Weight Support Treadmill on Cardiopulmonary Exercise Capacity and Trainability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AlterG-Training-I Studie
Record Dates: First submitted 2016-10-12; First posted 2016-11-01 (Estimated); Last update posted 2022-05-25 (Actual); Status verified 2021-09

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AlterG Anti-gravity treadmill (Active Comparator): cont. aerobic exercise training with lower body weight support
  Interventions: Other: AlterG Anti-gravity treadmill
- Exercise without body weight support (No Intervention): cont. aerobic exercise training without lower body weight support

INTERVENTIONS:
Other: AlterG Anti-gravity treadmill — Participants in this group will complete a 12 week aerobic exercise training protocol with 40% lower body weight support on an AlterG Anti-gravity treadmill
  Arms: AlterG Anti-gravity treadmill

SUMMARY:
The AlterG®-anti-gravity treadmill provides lower body weight support which enables individuals to exercise without feeling their full body weight. How this body weight support influences cardiovascular, respiratory, vascular and metabolic parameters is currently unclear. Further, whether body weight support influences the trainability in response to moderate continuous exercise is unknown. This investigation has two main goals. First, we explore the direct influence of lower body weight support on cardiometabolic parameters during maximal exercise testing. Second, we aim to compare changes in cardiorespiratory fitness in response to a structured exercise protocol using moderate intensity with and without lower body weight support.

ELIGIBILITY:
Inclusion Criteria:

* maximal oxygen consumption below age-sex specific standard

Exclusion Criteria:

* acute infection within the last four weeks
* anemia (males: Hb < 8.1 mmol/L; females Hb < 7.4 mmol/L)
* previous reports of myo-, endo, or pericarditis
* previous stroke or acute myocardial infarction
* heart failure (NYHA > 1)
* aortic valve stenosis
* congenital heart disease
* cardiomyopathy
* severe left ventricular hypertrophy
* cardiac arrythmias
* hypertension
* diabetes
* BMI > 35
* cancer
* pregnancy
* aneurysm of aorta or cerebral arteries

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Maximal oxygen consumption | 12 weeks
  VO2peak [ml/min]

SECONDARY OUTCOMES:
Oxygen consumption at anaerobic threshold | 12 weeks
  VO2@AT
Pulse wave velocity | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Dörr, M.D., Principal Investigator — University Medicine Greifswald
Locations (1):
- Cardiovascular examination center of the University Medicine Greifswald, Greifswald, Germany

REFERENCES:
- [Derived] Brussau T, Oehring R, Felix SB, Dorr M, Bahls M. Cardiorespiratory and metabolic responses to exercise testing during lower-body positive pressure running. J Appl Physiol (1985). 2020 Apr 1;128(4):778-784. doi: 10.1152/japplphysiol.00328.2019. Epub 2020 Feb 13. PMID 32053417